CLINICAL TRIAL: NCT03754348
Title: Microglial Activation in Narcolepsy Type 1 and Kleine-Levin Syndrome: Positron Emission Tomography (PET) Study in [18F] DPA-714
Acronym: NARCOGLIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RECHMPL18_0067
Record Dates: First submitted 2018-11-05; First posted 2018-11-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2022-03

CONDITIONS: Narcolepsy 1; Kleine-Levin Syndrome
Keywords: narcolepsy type 1; orexin; hypocretin; [18F] DPA-714; biomarker; auto immunity; kleine-levin syndrome
MeSH Terms: conditions — Narcolepsy 1; Kleine-Levin Syndrome | interventions — Magnetic Resonance Spectroscopy; Product Labeling; N,N-diethyl-2-(2-(4-(2-fluoroethoxy)phenyl)-5,7-dimethylpyrazolo(1,5-a)pyrimidin-3-yl)acetamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NT1 group (Experimental): hypothalamus neuroinflammation evaluation in Narcoleptic patients
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714
- Control group (Other): hypothalamus neuroinflammation evaluation in control patients (patients without hypersomnia or inflammatory pathology)
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714
- KLS group (Experimental): hypothalamus neuroinflammation evaluation in Kleine-Levin syndrome patients
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714

INTERVENTIONS:
Radiation: PET scan with tracer injection [18F] DPA-714 — the subject will receive a dose of 3.5MBq / kg intravenous (in bolus) more or less 20%, knowing that the minimum dose injected is unchanged at 150MBq and the maximum dose at 370 MBq. Irradiation will remain below 10 mSv

SUMMARY:
Type 1 narcolepsy (NT1) is a chronic sleep disorder caused by the selective and irreversible loss of neurons from the hypothalamus, which synthesizes a neurotransmitter: hypocretin (Hcrt) / orexin. The exact cause of this destruction is still unknown, but the autoimmune hypothesis is strongly favored, involving the interaction of genetic and environmental factors. The treatment of NT1 is currently only symptomatic, targeting hypersomnolence and cataplexy. To prevent the destruction of Hcrt neurons, immunomodulatory agents have been tested, with varying efficacy, probably due to varying degrees of hypothalamic impairment and stages of disease progression. During microglial activation, a condition associated with neuroinflammation in the brain, there is an increase in the mitochondrial translocation protein (TSPO), which can be quantified in vivo by specific tracers, such as the [18F] DPA- 714, in positron emission tomography (PET), a very sensitive nuclear imaging technique. The aim here is to study microglial activation in PET [18F] DPA-714 in NT1 patients with recent evolution in comparison with controls; then analyze the effect of age, and the severity of symptoms on this PET imaging biomarker. The hypothesis is that microglial activation, especially of the hypothalamic region, is greater in NT1 than controls.

DETAILED DESCRIPTION:
Formerly known as narcolepsy with cataplexy, narcolepsy type 1 (NT1) is a rare and disabling sleep pathology that affects 0.02% of the population. It occurs mainly in young adults and children, with repercussions throughout their existence. It is characterized by excessive daytime sleepiness (EDS), which is often the most disabling symptom. Diurnal sleep access is irrepressible, typically short-lived, and refreshing. Cataplexies are the most specific, almost pathognomonic sign of this condition. It is a loss of muscle tone in full consciousness, sudden, triggered by an often positive emotion (laugh, excitement, joke). Nighttime sleep is also disturbed and there may be other signs of paradoxical sleep dysregulation such as hypnagogic hallucinations (at sleep) or hypnopompic (waking) hallucinations, and sleep paralysis.

The diagnosis is confirmed by a polysomnographic recording (PSG) followed by iterative sleep latency tests (TILE) the next day. According to the new international criteria (ICSD-3), patients have a sleep latency of less than or equal to 8 minutes to TILE, and at least 2 sleep in paradoxical sleep (ESP) . An ESP during the previous night PSG can replace a TILE ESP. Typical cataplexies must also be found during the interrogation, but a level of hypocretin-1 collapsed in cerebrospinal fluid (CSF) (<110 ng / L) can now be sufficient for diagnosis, given its very high specificity ( 99%) and sensitivity (> 87%) for NT1.

NT1 is due to the selective and irreversible loss of Hcrt neurons. The exact cause of this destruction is still unknown, but the autoimmune hypothesis is strongly favored. The etiology is probably multifactorial, involving genetic and environmental factors. In fact, 97% of patients with NT1 are carriers of the HLA (Human Leukocyte Antigen) allele DQB1 * 06: 02, a class II major histocompatibility complex (MHC) allele.

Treatments of NT1 are currently only symptomatic, targeting the different symptoms: drowsiness, poor sleep at night, cataplexy, and other symptoms related to dysregulation of sleep Microglial activation is involved in the neuroinflammation process of certain central nervous system pathologies.

When microglia are activated, following aggression or cellular inflammation, the expression of TSPO increases. Positron Emission Tomography (PET) is a nuclear imaging technique that can be used to create anatomical and molecular images with high sensitivity. New TSPO-specific tracers have been recently developed, such as [18F] DPA-714, to quantify in vivo microglial activation in brain PET.

The goal here is to study the cerebral microglial activation in PET in NT1 patients with recent evolution (appearance of the first symptoms - somnolence and cataplexy - less than 2 years ago) in comparison with controls; then analyze the effect of age, and the severity of symptoms on this PET imaging biomarker. Thus, we hypothesize microglial activation, particularly of the hypothalamic region, in NT1 patients at an early stage of disease progression, possibly correlated with the severity of symptoms. To test this hypothesis, we will compare the in vivo microglial activation with PET [18F] DPA-714 in NT1 subjects, versus control subjects followed for another age-and-sex-matched non-narcolepsy and hypersomnia-free sleep pathology. The images will be analyzed semi-quantitatively by determining SuVr (or normalized binding value), a method validated in international studies.

ELIGIBILITY:
Inclusion criteria:

1. For all groups :

   * Written agreement for participation
   * Able to understand instructions and information data
   * Without any immunomodulatory, immunosuppressant, or anti-inflamatory medication
2. For NT1 patients:

   * 10 years-old or more
   * Responding to NT1 criteria (ICSD-3)
   * Under psychostimulant or not for narcolepsy
3. For KLS patients:

   * 10 years-old or more
   * KLS diagnosis
4. For controls

   * 18 years-old or more
   * Absence of narcolepsy
   * Absence of acute or chronic inflammatory disease

Exclusion criteria (for all groups):

* People without public insurance regime
* Specific contraindication to the use of PET (specific allergy related to the ligand).
* Pregnant and breastfeeding women
* Persons deprived of liberty by judicial or administrative decision
* People hospitalized without consent, or subject to legal protection
* Persons unable to consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Quantification of microglial activation in the hypothalamus (SuVr) of adult NT1 patients compared to controls | 1 day

SECONDARY OUTCOMES:
Correlation between microglial activation in the hypothalamus, thalamus, and other regions of interest in adult and child patients and severity of the disease | 1 day
Correlation between microglial activation in the hypothalamus, thalamus, and other regions of interest in adult and child patients and electrophysiological biomarkers | 1 day
Correlation between microglial activation in the hypothalamus, thalamus, and other regions of interest in adult and child patients and inflammatory biomarkers | 1 day
Microglial activation in the hypothalamus, thalamus, and other regions of interest in KLS patients vs NT1 patients | 1 day
Correlation between microglial activation in the hypothalamus, thalamus, and other regions of interest in KLS patients and time and severity of the disease (clinical, polysomnographic and biologic parameters) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

REFERENCES:
- [Derived] Barateau L, Krache A, Da Costa A, Lecendreux M, Debs R, Chenini S, Arlicot N, Vourc'h P, Evangelista E, Alonso M, Salabert AS, Silva S, Beziat S, Jaussent I, Mariano-Goulart D, Payoux P, Dauvilliers Y. Microglia Density and Its Association With Disease Duration, Severity, and Orexin Levels in Patients With Narcolepsy Type 1. Neurology. 2024 May;102(10):e209326. doi: 10.1212/WNL.0000000000209326. Epub 2024 Apr 26. PMID 38669634